CLINICAL TRIAL: NCT00121316
Title: Safety and Efficacy of Pimecrolimus Cream 1% in Mild to Moderate Head and Neck Atopic Dermatitis (AD) of Patients Intolerant to, or Dependant on, Topical Corticosteroids
Brief Title: Safety and Efficacy of Pimecrolimus Cream 1% in Mild to Moderate Head and Neck Atopic Dermatitis (AD) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CASM981C2442
Record Dates: First submitted 2005-07-13; First posted 2005-07-21 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; pimecrolimus
MeSH Terms: conditions — Dermatitis, Atopic | interventions — pimecrolimus

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Pimecrolimus
  Interventions: Drug: Pimecrolimus
- 2 (Placebo Comparator): Matching vehicle cream (placebo)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pimecrolimus — Pimecrolimus Cream 1 %
  Other Names: Elidel
  Arms: 1
Drug: Placebo — Vehicle cream (placebo cream)
  Arms: 2

SUMMARY:
This study is not being conducted in the United States.

Patients who are intolerant of topical corticosteroids (TCS) have either experienced an adverse event resulting from the use of TCS, or require unacceptable levels of exposure to TCS in order to control their AD. This is of particular concern for patients with recurrent flares on delicate skin areas such as the head and neck.

The purpose of this study is to investigate whether pimecrolimus cream 1%, a non-steroidal anti-inflammatory drug, is efficacious in treating mild to moderate head and neck AD in patients who are intolerant of, or dependent on topical corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* 12 years of age or older
* Mild to moderate facial AD at screening (facial IGA 2 - 3)
* Patients intolerant of, or dependent on, topical corticosteroids
* Diagnosis of atopic dermatitis by the Hanifin and Rajka criteria
* For female patients, a negative pregnancy test. Women who are pregnant or who are breast-feeding may not be included in the study. Women of child-bearing potential must follow a medically recognized form of contraception.

Exclusion Criteria:

At baseline and throughout the study, patients:

* Who have AD on greater than 30% of total body surface area in addition to facial eczema
* Who have concurrent skin disease (e.g. acne) in the study area or active skin infections (active bacterial, viral or fungal infections or infestations, herpes simplex, herpes zoster, chicken pox), or other conditions that may interfere with the evaluation (e.g. generalized erythroderma, Netherton's syndrome)
* Who are immunocompromised (e.g. Lymphoma, AIDS, Wiskott-Aldrich Syndrome) or have a history of malignant disease (with the exception of treated basal-cell carcinoma)
* Who have previously reported poor, no clinical response, or hypersensitivity to topical pimecrolimus cream (Elidel)
* Who have received phototherapy (e.g. UVA, UVB) or systemic therapy (e.g.immunosuppressants, corticosteroids, cytostatics) known or suspected to have an effect on AD within 4 weeks of Visit 2
* Who have received investigational drugs within 8 weeks of first application of study drug or planned use of other investigational drugs during participation of this study
* Who are unlikely to comply with therapy

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2004-10; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
The percentage of patients who have a facial Investigator's Global Assessment (IGA) score of 0 or 1 (clear or almost clear)

SECONDARY OUTCOMES:
Percentage of responders in overall Eczema Area and Severity Index (EASI) score
Percentage of responders in the head and neck EASI score
Percentage of patients achieving at least a 60 % reduction from baseline in the head and neck EASI score
Percentage of patients achieving a score of 0 or 1 for the pruritus score (absent or mild)
Effects on skin atrophy and telangiectasia (spider veins) existing at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (1):
- This study is not being conducted in the United States, Novartis Pharma AG, Switzerland